CLINICAL TRIAL: NCT04770090
Title: Preliminary Descriptive Exploratory Pilot Study Research of Circulating Tumor Cells Released During Cervical Cancer Surgery
Brief Title: Research of Circulating Tumor Cells Released During Cervical Cancer Surgery
Acronym: CTC-COL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other); Institut du Cancer de Montpellier - Val d'Aurelle (Other); Laboratoire Cellules Circulantes Rares Humaines (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL20_0090
Record Dates: First submitted 2021-02-04; First posted 2021-02-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer Stage IA1; Cervical Cancer Stage IB1; Cervical Cancer Stage IA2; Cervical Cancer Stage IB2
Keywords: Cervical cancer; Circulating tumor cell; Coelioscopy; Disease-free survival; Laparoscopy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Early stage cervical cancer (Experimental): Patients with cervical cancer eligible for surgery, stage IA1 to IB2
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Peripheral blood samples at the beginning of surgery, after pneumoperitoneum creation and uterine pedicles coagulation.

SUMMARY:
Cervical cancer is a rare pathology. Recent studies showed that the risk of recurrence is higher for patients treated by coelioscopy in comparison with laparotomy. It could be explained by the spread of circulating tumor cells (CTC) due to tumor mobilization during different steps of the surgery.

The primary goal is to evaluate the spread of CTC during surgery on peripheral blood samples.

The secondary outcome is to evaluation the disease-free survival at 3 and 5 years postoperatively.

20 patients with early stage cervical (IA1 to IB2) eligible to coelioscopic stadification and laparoscopic surgery will be included.

DETAILED DESCRIPTION:
CTC detection could be a pronostic factor for cancer evolution. Cervical cancer is a rare pathology with increased death rate.

Despite recommendations for coelioscopic treatment of < 4cm cervical cancers, recent studies showed that the risk of recurrence is higher for patients treated by coelioscopy in comparison with laparotomy. It could be explained by the spread of circulating tumor cells (CTC) due to tumor mobilization during coelioscopic stadification and laparoscopic surgery.

Hypothesis : Mobilization of the tumor during coelioscopy leads to CTC spread. This spread could explain the recurrence of cervical cancer.

This pilot study will evaluate the possibility of CTC detection during surgery. The primary goal is to evaluate the spread of CTC during the different steps of surgery on peripheral blood samples.

The secondary outcome is to evaluation the disease-free survival at 3 and 5 years postoperatively.

20 patients with early stage cervical (IA1 to IB2) eligible to coelioscopic stadification and laparoscopic surgery will be included.

ELIGIBILITY:
Inclusion Criteria:

* Woman >18 years old
* Cervical cancer confirmed by histology
* Early stage eligible for immediate surgical treatment (or post-brachytherapy): stages IA1, 1A2, 1B1 and IB2 with or without emboli determined by MRI performed as part of the treatment
* Histology : epidermoid carcinoma and adenocarcinoma
* Valid Social Security
* Wrote consent

Exclusion Criteria:

* Advanced stage (Stage IB3 and more)
* Concomitant cancer
* Pregnant or breastfeeding woman
* Vulnerable person (Article L1121-6 of the Public Health Code)
* Participation to other study with an exclusion period still in progress
* Participation to other study that may have an impact on the prognosis of cervical cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Number of circulating tumor cell detected after cervical cancer surgery. | Within 48 hours after surgery.
  Detection of the presence of at least one circulating tumor cell from blood samples taken during surgery (one CTC per 7.5mL of blood or increase of at least one CTC if CTC is present pre-operatively)

SECONDARY OUTCOMES:
Evaluation of disease-free survival | Two points at the 3rd and 5th years
  The disease-free survival will be evaluated at 3 and 5 years post-operatively

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Department of gynaecology, Montpellier University Hospital, Montpellier
  - Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier
  - CHU de Nîmes, Nîmes

IPD SHARING:
Plan to Share IPD: No